CLINICAL TRIAL: NCT04091204
Title: A Phase II Trial of Olaparib in Patients With Recurrent Ovarian Cancer Wild Type for Germline and Somatic BRCA 1 and 2 Genes: The MITO 31 Translational Study
Brief Title: Olaparib in Patients With Recurrent Ovarian Cancer Wild Type for Germline and Somatic BRCA 1 and 2 Genes: The MITO 31 Translational Study
Acronym: MITO 31
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MITO 31; 2018-000617-20 (EudraCT Number)
Record Dates: First submitted 2019-09-09; First posted 2019-09-16 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: BRCA Wild Type Platinum Sensitive Recurrent Ovarian Cancer
Keywords: wild-type BRCA 1 and 2; platinum sensitive; recurrent ovarian cancer; olaparib; maintenance treatment
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib

STUDY DESIGN:
Intervention Model Description: This is a single arm, multicentre, open-label Phase 2 study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Olaparib (Experimental): Olaparib is given orally at the dose of 300 mg bid continually as maintenance therapy after a platinum based chemotherapy
  Interventions: Drug: Olaparib tablets

INTERVENTIONS:
Drug: Olaparib tablets — Olaparib is given orally at the dose of 300 mg bid continually as maintenance therapy after a platinum based chemotherapy

SUMMARY:
The aim of the study is to explore a prognostic clinical and molecular biomarker profile in a population of BRCA wild-type recurrent high-grade ovarian cancer patients treated with olaparib as maintenance after response to a platinum based therapy as platinum sensitive recurrence treatment.

DETAILED DESCRIPTION:
This is a single arm, open-label Phase 2 study designed to evaluate the effect of maintenance olaparib treatment after response to platinum-based chemotherapy in patients with BRCA wild type platinum sensitive recurrent ovarian cancer. The goal is to identify a clinical and molecular profile able to select a group of patients, treated with olaparib as maintenance, with a favorable prognosis.

ELIGIBILITY:
Inclusion Criteria

1. Patients must be ≥ 18 years of age
2. Female patients with histologically diagnosed relapsed high grade ovarian cancer (including primary peritoneal and /or fallopian tube cancer)
3. Documented absence of somatic and germline mutations of BRCA1 or BRCA2 genes, that is predicted to be deleterious or suspected deleterious
4. ECOG Performance Status of 0-2
5. Patients must have a life expectancy of at least 16 weeks
6. Signed informed consent obtained prior to initiation of any study-specific procedures and treatment as confirmation of the patient's awareness and willingness to comply with the study requirements
7. Availability of tumor and blood samples for molecular analyses
8. Patients who have received at least 2 previous line of platinum containing therapy prior to randomization

   * For the penultimate chemotherapy course prior to enrolment on the study:
   * Patient defined as platinum sensitive after this treatment, defined as having disease progression greater than 6 months after completion of their last dose of platinum chemotherapy

For the last chemotherapy course immediately prior to randomization on the study:

* Patients must be, in the opinion of the investigator, in radiologic response (partial or complete response) according to RECIST 1.1 criteria, or may have no evidence of disease (if optimal cytoreductive surgery was conducted prior to chemotherapy), and no evidence of a rising CA-125 compared to nadir value, following completion of this chemotherapy course i. Patient must have received, at least 4 cycles of a platinum based chemotherapy regimen (e.g. carboplatin or cisplatin per standard clinical practice) j. Patients must be enrolled within 8 weeks of their last dose of chemotherapy k. Maintenance treatment, including bevacizumab, is allowed at the end of the penultimate platinum regimen l. Postmenopausal or evidence of non childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1 m. Patients must have normal organ and bone marrow function measured within 28 days prior to administration of study treatment as defined below:
* Hemoglobin ≥ 10.0 g/dL with no blood transfusion in the past 28 days
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 100 x 109/L
* Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (Serum Glutamic Oxaloacetic Transaminase (SGOT)/ Alanine aminotransferase (ALT) (Serum Glutamic Pyruvate Transaminase (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be ≤ 5x ULN
* Patients must have creatinine clearance estimated using the Cockcroft-Gault equation of ≥ 51 mL/min:

Estimated creatinine clearance= (140-age [years]) x weight (kg) (x F)a serum creatinine (mg/dL) x 72 a where F=0.85 for females and F=1 for males

Exclusion Criteria

1. History or evidence of synchronous primary endometrial carcinoma, unless all of the following criteria related to the endometrial carcinoma are met:

   * stage ≤ IA
   * no more than superficial myometrial invasion
   * no lymph vascular invasion
   * not poorly differentiated (grade 3 or papillary serous or clear cell carcinoma)
2. Other malignancy within the last 5 years, except for adequately treated non melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinomna in situ (DCIS), stage 1, grade 1 endometrial carcinoma, or other solid tumours including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for > 5years
3. Resting ECG with QTc > 470 msec on 2 or more time points within a 24 hour period or family history of long QT syndrome
4. Participation in another clinical study with an investigational product during the chemotherapy course immediately prior to randomization
5. Patients receiving any systemic radiotherapy (except for palliative reasons) within 3 weeks prior to study treatment
6. Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting olaparib is 2 weeks
7. Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort ) or moderate CYP3A inducers (eg. bosentan, efavirenz, modafinil). The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents
8. Persistent toxicities [>Common Terminology Criteria for Adverse Event (CTCAE) grade 2)] caused by previous cancer therapy, excluding alopecia
9. Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML
10. Patients with symptomatic uncontrolled brain metastases. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study as long as these were started at least 4 weeks prior to treatment
11. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days
12. Major surgery within 2 weeks of starting study treatment and patients must have recovered from any effects of any major surgery
13. Patients considered at poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on High Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent
14. Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
15. Breast-feeding women
16. Immunocompromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV)
17. Patients with a known hypersensitivity to olaparib or any of the excipients of the product
18. Patients with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids
19. Previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
20. Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable)
21. Any previous treatment with PARP inhibitor, including olaparib
22. Involvement in the planning and/ or conduct of the study
23. Previous enrolment in the present study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients with histologically diagnosed relapsed high grade ovarian cancer (including primary peritoneal and /or fallopian tube cancer)
Enrollment: 200 (Estimated)
Dates: Start 2019-07-04 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | up to 24 months
  as determined by investigator

SECONDARY OUTCOMES:
Overall Survival | up to 36 months
  as determined by investigator
Progression Free Survival 2 | up to 36 months
  as determined by investigator, after the subsequent line of treatment
Worst grade toxicity per patient | evaluated at each cycle every 28 days (during maintenance therapy), up to 30 days after cessation of olaparib
  graded according to Common Terminology Criteria for Adverse Event (CTCAE) version 5.0
Response Rate | up to 24 months
  according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Pignata, MD, PhD, Principal Investigator — National Cancer Institute, Naples; Clorinda Schettino, MD, Study Chair — National Cancer Institute, Naples; Francesco Perrone, MD, PhD, Study Chair — National Cancer Institute, Naples
Locations (1):
- Istituto Nazionale dei Tumori , Oncologia Medica - Dipartimento Uro-Ginecologico, Napoli, Italy

IPD SHARING:
Plan to Share IPD: No